CLINICAL TRIAL: NCT03256292
Title: Long-term Lifestyle Change in Obese Older Veterans
Brief Title: Long-term Lifestyle Change and Testosterone Replacement
Acronym: LITE
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Dennis T. Villareal, Professor, Baylor College of Medicine
Other Study IDs: H-40598
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Hypogonadism; Aging; Overweight and Obesity
MeSH Terms: conditions — Hypogonadism; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- testosterone, diet, and increased physical activity: Group receiving standard of care consisting of diet and regular exercise counseling + testosterone replacement therapy
  Interventions: Drug: Testosterone replacement; Behavioral: lifestyle

INTERVENTIONS:
Drug: Testosterone replacement — Testosterone replacement therapy
Behavioral: lifestyle — lifestyle intervention consisting of diet and increased physical activity

SUMMARY:
Older hypogonadal obese veterans previously participated in a 6 month lifestyle change (diet-induced weight loss and exercise) study with or without testosterone replacement therapy before being followed for the following year at the clinic while receiving standard of care consisting of diet and exercise counseling (for healthy lifestyle change) and testosterone replacement therapy. This study will determine if long-term lifestyle change and testosterone replacement therapy with associated improvement in physical and metabolic health can be maintained in obese older adults.

DETAILED DESCRIPTION:
Background: There are studies on long-term testosterone replacement in older adults with hypogonadism showing benefits on body composition, sexual function and mood but not on testosterone replacement therapy in combination with lifestyle change (diet-induced weight loss and exercise) in the specific population of older adults with both obesity and hypogonadism.

Purpose: To determine if long-term lifestyle change and testosterone replacement therapy with associated improvement in physical and metabolic health can be maintained in obese older adults .

Design: Overweight/obese older veteran patients with obesity and hypogonadism who are being followed at the endocrine clinic while receiving standard of care consisting of diet and exercise counseling (for healthy lifestyle change) and testosterone replacement therapy will be recruited for testing of physical, metabolic, cognitive/mood, quality of life, and body composition testing.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese (BMI = or > 27 kg/m2)
* Older (65-85 yr)
* Male veteran patients being seen at the PI's endocrine clinic and receiving standard of care consisting of diet and regular exercise counseling
* Diagnosed with hypogonadism on current or previous testosterone replacement at the PI's endocrine clinic
* Willing to provide informed consent

Exclusion Criteria:

* Failure to provide informed consent
* Unstable cardiopulmonary disease (e.g. recent MI, unstable angina, stroke) or unstable disease (Class III or IV congestive heart failure).

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults with hypogonadism following lifestyle change (diet and exercise on their own for at least one year) with testosterone replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Physical Performance Test score | 18 month
  The primary functional outcome is the modified physical performance test, which includes seven standardized tasks (walking 50 ft, putting on and removing a coat, picking up a penny, standing up from a chair, lifting a book, climbing one flight of stairs, and performing a progressive Romberg tests) plus two additional tasks (climbing up and down four flights of stairs and performing a 360-degree turn). The score for each task ranges form 0 to 4; a perfect score is 36.
Change in body weight | 18 month
  Measured after an overnight fast using calibrated scales

SECONDARY OUTCOMES:
Change in body composition (lean mass, fat mass and bone mineral density) | 18 month
  Assessed by using dual-energy x-ray absorptiometry
Volumetric BMD | 18 month
  Assessed by using peripheral quantitative computed tomography (pQCT)
Biochemical Markers of Bone Turnover (Serum C-terminal telopeptide (CTX) | 18 month
  measured by ELISA
Change in prostate specific antigen | 18 month
  measured in the blood
Prostate Symptom Assessment | 18 month
  Using the International Prostate Symptom Scoring
Mood | 18 month
  Using the Geriatric Depression Scale
Quality of Life | 18 month
  Using SF-36 and impact of weight on quality of life short form (IWQOL-lite)
Sexual function | 18 month
  Using the International Index of Erectile Function
Change in trabecular bone score | 18 month
  Using DXA
Change in muscle strength and quality | 18 month
  Using biodex dynamometry
Change in balance | 18 month
  as measured by leg stance and obstacle course
Change in Functional Status | 18 month
  Using functional status questionnaire
Change in gait | 18 month
  as measured by completing the time to walk a certain distance
Change in bone quality | 18 month
  Using HrpQCT
Change in testosterone level | 18 month
  as measured in the blood
Change in sex hormone globulin | 18 month
  as measured in the blood
Change in metabolic hormones | 18 month
  Leptin, adiponectin, and similar metabolic hormones as measured in the blood
Change in Composite cognitive z-score | 18 month
  using cognitive instrument testing
Change in Modified mini-mental exam | 18 month
  using cognitive instrument testing
Change in Stroop color naming | 18 month
  using cognitive instrument testing
Change in Word list fluency | 18 month
  using cognitive instrument testing
Change in Ray auditory verbal learning test | 18 month
  using cognitive instrument testing
Change in Trail A/B | 18 month
  using cognitive instrument testing
Change in waist circumference | 18 month
  as measured
Change in serum PTH | 18 month
  as measured in the blood
Change in lipid profile | 18 month
  as measured in the blood
Change in blood pressure | 18 month
  as measured by sphygmomanometry
Change in metabolic syndrome | 18 month
  using harmonized metabolic syndrome criteria
bone strength index | 18 months
  assessed by pQCT
Cortical to total area | 18 months
  assessed by pQCT
Change in density weighted polar section modulus | 18 months
  assessed by pQCT
Change in cortical density | 18 months
  assessed by pQCT
Change in cortical area | 18 months
  assessed by pQCT
Change in Biochemical Markers of Bone Turnover (PINP) | 18 months
  measured by RIA
Change in lipid profile | 18 months
  measured in the blood
Change in vitamin D level | 18 months
  measured in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Villareal, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
A De-identified, Anonymized Dataset will be created and shared. NOTE: ORO recommends that such sharing take place under a written agreement that adheres to any applicable Informed Consent provisions and prohibits the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. However, it is permissible for final datasets in machine-readable format to be submitted to and accessed from PubMed Central (and similar sites) provided that care is taken to ensure that the individuals cannot be re-identified using other publicly available information.
Supporting Information: Study Protocol
Time Frame: Controlled access requests will be provided to the greatest extent possible under specific DUAs or other written agreements and open access will be provided to the final datasets underlying peer-reviewed publications in accordance with the research disposition policy which states that research records will be destroyed 6 years after cutoff (at the end of the fiscal year) after completion of the research project, but may be retained longer if required by other federal regulations or sponsor archive requirements.
Access Criteria: Controlled access requests will be provided to the greatest extent possible under specific DUAs or other written agreements and open access will be provided to the final datasets underlying peer-reviewed publications in accordance with the research disposition policy which states that research records will be destroyed 6 years after cutoff (at the end of the fiscal year) after completion of the research project, but may be retained longer if required by other federal regulations or sponsor archive requirements.